CLINICAL TRIAL: NCT05879315
Title: Stratification of Fall Risk in a Rehabilitation Department Through Tools That Evaluate Postural Balance and Movement Capacity in the Preoperative Period
Brief Title: Evaluation of Balance and Movement in Order to Prevent the Risk of Falling in the Post-operative Period
Acronym: NOCADINRIAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CE AVEC: 888/2022/Sper/IOR
Record Dates: First submitted 2023-03-14; First posted 2023-05-30 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Patient Fall
MeSH Terms: interventions — Hospitals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- risk stratification of fall in patients waiting for hip and knee surgery (Other)
  Interventions: Other: Fall risk prevention in hospital

INTERVENTIONS:
Other: Fall risk prevention in hospital — All patients (hip and knee) upon admission to the Orthopedic Department of the DRS (Rizzoli Sicily Department), throughin the pre-operative setting will undergo an assessment of mobility level, dynamic stability and co-ordination: Test UP and GO, Il Four Square Step Test, Stabilometric Analysis. After admission to the DRS Rehabilitation Medicine Department, hip and knee will receive an evaluation, which is currently used, consisting of: History of fall risk through multidimensional assessment, Compilation of ICF(International Classification of Functioning, Disability and Health) and Barthel Index. The following ratings will also be added: Compiling the Morse scale, Pharmacological history, CIRS (Cumulative Illness Rating Scale)

SUMMARY:
This study aims to identify, in patients undergoing hip and knee joint replacement, the functional evaluation tools predictive of the risk of falling upon admission to the orthopedic department and to correlate the results obtained with clinical evaluation scales that are generally used for fall risk stratification and the number of falls actually occurring both in the orthopedic department and in the rehabilitation department.

DETAILED DESCRIPTION:
The goal of this prospective interventional cohort study is to identify functional assessment tools predictive of the risk of falling in patients undergoing hip and knee joint replacement surgery upon admission to an orthopedic department and to correlate the results obtained with the clinical rating scales generally used for the risk stratification of fall. All patients upon admission to the Orthopedic Department of the DRS (Rizzoli Sicily Department), throughin the pre-operative setting will undergo an assessment of mobility level, dynamic stability and co-ordination: Test UP and GO, Il Four Square Step Test, Stabilometric Analysis. After admission to the DRS Rehabilitation Medicine Department, all patients will receive an evaluation, which is currently used, consisting of: History of fall risk through multidimensional assessment, Compilation of ICF(International Classification of Functioning, Disability and Health) and Barthel Index. The following ratings will also be added: Compiling the Morse scale, Pharmacological history, CIRS (Cumulative Illness Rating Scale), The scores obtained from the various measures used in the patients will be correlated to any falls recorded during hospitalization with the aim to obtain a stratification of falls risk in those patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient's ability to perform the required tests, the understanding of the language of the study
* Patients of both sexes between the ages of 50 and 85;
* Patients candidates for hip and knee joint replacement in the Orthopedic Department of the DRS.

Exclusion Criteria:

* Non-ambulatory patients, patients with amputation of one of the 2 lower limbs,
* Serious neurological and/or psychiatric diseases
* Patients with vestibular deficits

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Test UP and GO. The time of performance is measured in seconds and lower values indicate better balance control and lower fall risk. | Just Baseline
  Participants have been instructed to get up from a chair, walk up to a sign marked on the floor 3 meter ahead on the chair, turn around in their own circles, walk up to the chair and sit down. The time of performance is measured in seconds and lower values indicate better balance control and lower fall risk.
Four Square Step Test. The time of performance is measured in seconds | Just Baseline
  This test evaluates the dynamic balance of patients. The test involves the execution of a pre-established series of steps (forward, lateral, backward) within four squares. The time taken to complete one clockwise and one counterclockwise revolution is taken as a reference parameter.
  The 15-second threshold helps us assess the risk of falling in the population being studied.
  Times longer than 15 seconds are associated with a higher risk of falling. The young population is around 6-7 seconds.
Barthel Index. It is a questionnaire | Just Baseline
  The index, has it to establish the patient's degree of independence. It is made up of 10 items that include the municipalities daily activities (ADL Activities of Daily Living). Each item is assigned a score, the sum (maximum 100) indicates the degree of autonomy of the patient in carrying out the activities of daily life, the higher the score, the greater the autonomy of the subject.
Cumulative Illness Rating Scale. The scale has a cumulative score, which can range from 0 to 56 | Just Baseline
  It is a standardized tool used in the medical field to measure the patient's health as objectively as possible. The tool is clinical in nature and requires the physician to evaluate and measure the clinical and functional severity of 14 categories of disease. For each of these pathologies a severity value must be defined, based on the clinical history, the physical examination and the symptoms declared by the patient. The scale has a cumulative score, which can range from 0 to 56. According to its developers, the maximum score is not compatible with the patient's life.
Stabilometric Test | Just Baseline
  The posturographic analysis has been led by stabilometric platform. The partecipations underwent a static analysis (stabilometric examina-tion) maintaining standing position with feet placed together with an angle of 30 grades between right and left heels at 2 cm of distance, firstly with open eyes for 51.2 seconds and after that with closed eyes for 51.2 seconds too, in order to analyse the time and frequency of oscillations and self-adjustments of the patient excluding the visual input.
Morse Scale. It is a questionnaire. | Just Baseline
  The Morse scale is a quick and easy way to assess a patient's likelihood of falling. The questions in the questionnaire should be addressed to the patient or, if there are physical and cognitive problems that prevent him from responding to a family member. It is a scale composed of 6 items: (i) history of falls, (ii) presence of pathologies at risk, (iii) outpatient aids, (iv) intravenous therapy, (v) type of gait and (vi) mental state". Each answer has a score.
  The sum of the scores obtained defines the risk of falling:
  0 to 24 = low risk 25 to 50 = medium risk equal to or > 51 = high risk
International classification of functioning, disability and health | Just Baseline
  The general function of the ICF classification is to provide a standard and unified language that serves as a reference model for the description of health and related states. It defines the components of health and some related components such as education and Work.
  The domains (= a practical and meaningful set of physiological functions, anatomical structures, actions, tasks, or related life areas) contained in the ICF can, therefore, be seen as domains of the health and related domains. These domains are described from a bodily, individual and social point of view in two lists main:
  1. Body functions and structures
  2. Activities and Participation
  The ICF is therefore no longer a classification of diseases (1980 version) but has instead become one classification of components of health.

CONTACTS AND LOCATIONS:
Overall Officials: serena rizzo, Principal Investigator — Rizzoli Orthopedic Institute
Locations (1):
- Rizzoli Orthopedic Institute, Bagheria, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No